CLINICAL TRIAL: NCT04670562
Title: Longitudinal Follow up of Patients With Pleural Effusion in South Korea
Brief Title: Longitudinal Follow up of Patients With Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-2006/618-311
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-04

CONDITIONS: Pleural Effusion, Malignant; Prognosis
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Pleural fluid samples and blood samples will be collected from each participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the clinical course of patients diagnosed with pleural effusion and determine various clinical factors and biomarkers associated that can predict the diagnosis and clinical outcome and prognosis of patients with pleural effusion due to specific causes.

DETAILED DESCRIPTION:
Patients who presented to Seoul National University Bundang Hospital with pleural effusion would be recruited. Pleural fluid and blood samples would be collected. All patients will receive routine diagnostic procedures and medical care and treatments according to the diagnosis; the original cancer if diagnosed with malignant effusion, and managements for pleural effusion control. Patients would be observed for the clinical course and prognosis up to 3 years without any interventions caused by this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with pleural effusion
* Patients who undergo thoracentesis and fluid analysis for diagnosis and management

Exclusion Criteria:

* Patients who refuse to be enrolled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who presented with pleural effusion and undergo diagnostic/therapeutic thoracentesis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | From date of diagnosis of malignant pleural effusion until the date of death, assessed up to 36 months.
  Mortality

SECONDARY OUTCOMES:
Disease progression | From date of diagnosis of malignant pleural effusion until the date of first documented disease progression, assessed up to 36 months.
  Progression of original malignancy or new metastasis occured

CONTACTS AND LOCATIONS:
Overall Officials: Yeon Wook Kim, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided